CLINICAL TRIAL: NCT02124200
Title: High Cessation Rates in Smokers Using Personal Vaporizers: A Prospective 6-month Pilot Study
Brief Title: High Cessation Rates in Smokers Using Personal Vaporizers
Acronym: VAPECIG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universita degli Studi di Catania (Other)
Responsible Party: Principal Investigator, Riccardo Polosa, Full Professor of Internal Medicine, Universita degli Studi di Catania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Personal Vape Pilot (Vapecig)
Record Dates: First submitted 2014-04-24; First posted 2014-04-28 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2014-06

CONDITIONS: Tobacco Addiction
MeSH Terms: interventions — Tobacco Use Cessation Devices

ARMS (1):
- EGO/CE4, 9mg nicotine (Other)
  Interventions: Device: EGO/CE4, 9mg nicotine

INTERVENTIONS:
Device: EGO/CE4, 9mg nicotine

SUMMARY:
E-cigarettes are proving to be an attractive long-term alternative to conventional cigarettes. Although they may also help smokers to remain abstinent during their quit attempt, recent clinical trials with first generation e-cigarettes have shown only modest quit rates. Second generation devices may result in much higher quit rates. Their efficacy and safety in long-term smoking cessation and/or smoking reduction studies have never been investigated.

In this prospective proof-of-concept study we monitored modifications in smoking habits of 50 regular smokers (unwilling to quit) who were asked to switch to a second generation device focusing on smoking reduction and smoking abstinence. Study participants were invited to attend a total of five study visits: at baseline, week-4, week-8, week-12 and week-24. Product usage, number of cigarettes smoked, and exhaled carbon monoxide (eCO) levels were measured at each visit. Smoking reduction and abstinence rates were calculated. Adverse events and participants' opinions of these products were also reviewed.

ELIGIBILITY:
Inclusion Criteria:Healthy smokers 18-60 years old, smoking ≥15 conventional cigarettes per day (cig/day) for at least 10 years were recruited using anti-smoking leaflets and by an approved kiosk located in the atrium of the university hospital (AOU 'Policlinico-V. Emanuele') promoting the smoking cessation services of the CPCT (Centro per la Prevenzione e Cura del Tabagismo, Università di Catania, Italy).

-

Exclusion Criteria:history of alcohol and illicit drug use, major depression or other psychiatric conditions. We also excluded subjects who reported recent myocardial infarction, angina pectoris, essential hypertension (>140mmHg systolic and/or >90mmHg diastolic), diabetes mellitus, severe allergies, poorly controlled asthma or other airways diseases

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-01; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
reducers | week-24 from baseline
  sustained 50% reduction in the number of cig/day at week-24 from baseline (reducers)

SECONDARY OUTCOMES:
heavy reducers and quitters | week-24 from baseline
  sustained 80% reduction in the number of cig/day (heavy reducers) and sustained smoking abstinence at week-24 (quitters)

CONTACTS AND LOCATIONS:
Locations (1):
- 1Centro per la Prevenzione e Cura del Tabagismo (CPCT), Azienda Ospedaliero-Universitaria "Policlinico-Vittorio Emanuele", Università di Catania,, Catania, Italy, Italy

REFERENCES:
- [Derived] Polosa R, Caponnetto P, Maglia M, Morjaria JB, Russo C. Success rates with nicotine personal vaporizers: a prospective 6-month pilot study of smokers not intending to quit. BMC Public Health. 2014 Nov 8;14:1159. doi: 10.1186/1471-2458-14-1159. PMID 25380748